CLINICAL TRIAL: NCT03682614
Title: Effect of Intrauterine Injection of Human Chorionic Gonadotropin Before Embryo Transfer on Clinical Pregnancy Outcome in Repeated Implantation Failure Patients With Normal Pathohistological Stage --Pilot Study
Brief Title: Effect of Intrauterine Injection of HCG on Clinical Pregnancy Outcome in Repeated Implantation Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P2018010
Record Dates: First submitted 2018-09-18; First posted 2018-09-24 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2019-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Culture Media

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCG group (Experimental): All patients will accept HCG 500IU intrauterine injection 2 days before blastocyte transfer
  Interventions: Drug: HCG
- control group (Placebo Comparator): All patients will accept same dose of culture medium intrauterine injection 2 days before blastocyte transfer
  Interventions: Other: culture medium

INTERVENTIONS:
Drug: HCG — we will use the catheter to pass through the cervix, and after that, the experiment Group will accept 40 μl 500 IU HCG injection into the uterine cavity 2 days before the blastocyst transfer.
  Arms: HCG group
Other: culture medium — The placebo group will accept 40 μl of culture medium injection into the uterine cavity 2 days before the blastocyst transfer.
  Arms: control group

SUMMARY:
Repeated implantation failure（RIF） is a insurmountable bottleneck in assisted reproductive technology, many studies have considered that the cause of two-thirds of implantation failure is the decreased endometrial receptivity. After exclude some major local immune factors(NK,CD138 cells) and implantation window out of phase, There are still a part of patients infertile .Human chorionic gonadotropin (hCG) is an early pre-implantation signal molecule secreted by the embryo, it can promote endometrial proliferation, increase blood flow and promote embryonic adhesion and inhibit self-regulated apoptosis of trophoblast cells. Previous studies showed that: intrauterine injection of HCG before embryo transfer can improve clinical outcomes in IVF/Intracytoplasmic sperm injection(ICSI). But some studies found that the intrauterine injection of HCG can not significantly improve the success rate of blastocyst transfer, and the reason may be the intrauterine injection of HCG time is too late to significantly increase the implantation rate. Would ahead of intrauterine injection of HCG be more effective? Thus, the patients of repeated implantation frozen embryo cycle according to the random principle accepted two kinds of transplants ways: ①intrauterine injection of HCG before blastocyst transfer; ②blastocyst transfer. Try to understand whether intrauterine injection of HCG can significantly improve the clinical pregnancy rate of blastocyst transfer in repeated implantation failure patients.

ELIGIBILITY:
Inclusion Criteria:

* repeated implantation failure patients: ≥ 3 times IVF-embryo transfer failed to help pregnancy (biochemical or non-pregnant)
* age ≤36 years old
* normal histopathological stage (+5-7)
* endometrial NK cell <4.5%
* 0 endometrial CD138 positive cell
* natural cycle frozen embryo transfer
* frozen blastocysts (≥4BC) embryos ≥ 1

Exclusion Criteria:

* Scar uterus (diverticulum or incision false lumen after cesarean section)
* intrauterine adhesions
* untreated hydrosalpinx
* adenomyosis (endometrial displacement)
* endometritis
* uterine fibroids compress the endometrium

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 28 days after blastocyst transfer

SECONDARY OUTCOMES:
clinical implantation rate | 28 days after blastocyst transfer
ongoing pregnancy rate | 70 days after blastocyst transfer
ectopic pregnancy rate | within 3 months after blastocyst transfer
abortion rate | within 28 weeks after blastocyst transfer

CONTACTS AND LOCATIONS:
Overall Officials: Fei Gong, Doctor, Principal Investigator — Reproductive and Genetic hospital of CITIC-xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China